CLINICAL TRIAL: NCT02076412
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Study of Fostamatinib Disodium in the Treatment of Persistent/Chronic Immune Thrombocytopenic Purpura
Brief Title: A Efficacy and Safety Study of Fostamatinib in the Treatment of Persistent/Chronic Immune Thrombocytopenic Purpura (ITP)
Acronym: FIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-935788-048; 2013-005453-76 (EudraCT Number)
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Immune Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fostamatinib Disodium (Experimental): Fostamatinib Disodium tablet 100 mg or 150 mg PO bid (morning and evening) over the course of 24 weeks.
  Interventions: Drug: Fostamatinib Disodium
- Placebo (Other): Placebo tablet PO bid (morning and evening) over the course of 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fostamatinib Disodium — Fostamatinib Disodium tablet 100 mg or 150 mg PO bid (morning and evening) over the course of 24 weeks.
  Other Names: R935788; R788; Fostamatinib
  Arms: Fostamatinib Disodium
Drug: Placebo — Placebo tablet PO bid (morning and evening)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether fostamatinib is safe and effective in the treatment of persistent/chronic Immune Thrombocytopenic Purpura (ITP).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of persistent/chronic ITP for at least 3 months
* Average platelet count< 30,000/µL (and none > 35,000 unless as a result of rescue therapy) from at least 3 qualifying counts

Exclusion Criteria:

* Clinical diagnosis of autoimmune hemolytic anemia
* Uncontrolled or poorly controlled hypertension
* History of coagulopathy including prothrombotic conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rigel Pharmaceuticals, Inc., Study Director — Rigel Pharmaceuticals,Inc.
Locations (35):
- Hematology Oncology Associates of Rockland Division of Highland Medical PC, Nyack, New York, United States
- Austria (3):
  - Medizinische Universitaet Wien / AKH Wien, Vienna, AU
  - Hanusch-Krankenhaus Wiener Gebietskrankenkasse, Vienna, AU
  - LKH Feldkirch at LKH Rankweil, Rankweil
- Bulgaria (4):
  - Specialized Hospital for Active Treatment of Hematology Diseases, EAD, Sofia, Department of Chemotherapy, Hemotherapy and Blood Inherited Diseases to Clinic of Clinical Hematology;, Sofia, BG
  - MHAT Hristo Botev, AD, Vratsa, First Internal Department, Vratsa, BG
  - UMHAT Dr. Georgi Stranski, EAD, Pleven, Clinic of Hematology, Pleven
  - UMHAT Aleksandrovska, EAD, Clinic of Clinical Hematology, Sofia
- Czechia (5):
  - Fakultni nemocnice Brno, Brno, CZ
  - Hospital Kyjov, Kyjov, CZ
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice, Linterní Klinika, Klinika hematologie, Prague
- Germany (5):
  - Universitaetsklinikum Giessen und Marburg (UKGM), Giessen, DE
  - Werlhof Institut GmbH, Hanover, DE
  - Charit Berlin - Campus Benjamin Franklin, Berlin
  - Marien Hospital Duesseldorf, Düsseldorf
  - Universittsklinikum Essen, Essen
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Sykehuset Østfold Fredrikstad, Fredrikstad
- Poland (8):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpital Uniwersytecki, Krakow
  - Wojewódzki Szpital Specjalistyczny im. M. Kopernika w Łodzi, Lodz
  - Specjalistyczny Gabinet Lekarski, Lublin
  - Szpital Wojewodzki w Opolu, Opole
  - Wojewodzki Szpital Specjalistyczny im. J. Korczaka, Słupsk
  - Instytut Hematologii I Transfuzjologii, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wrocrlaw, Wroclaw
- Romania (3):
  - Spitalul Clinic Judetean de Urgenta Tirgu-Mures, Sectia Medicina Interna 1, Compartiment Hematologie, Târgu Mureş, Mureș County
  - Spitalul Clinic Colentina, Hematologie, Bucharest
  - Spitalul Clinic Coltea, Hematologie, Bucharest
- Spain (4):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitariola Paz, Madrid
  - Hospital Universitari i Politécnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cooper N, Altomare I, Thomas MR, Nicolson PLR, Watson SP, Markovtsov V, Todd LK, Masuda E, Bussel JB. Assessment of thrombotic risk during long-term treatment of immune thrombocytopenia with fostamatinib. Ther Adv Hematol. 2021 Apr 30;12:20406207211010875. doi: 10.1177/20406207211010875. eCollection 2021. PMID 33995988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 74 patients were enrolled from January 2015 to August 2016
Groups:
- Fostamatinib Recipient: Fostamatinib (100 mg PO bid or 150 mg PO bid)
- Placebo Recipient: Placebo
Period: Overall Study
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Started | 50 | 24
Completed | 13 | 2
Not Completed | 37 | 22

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Fostamatinib Recipient | Placebo Recipient | Total
Number analyzed (Participants) | 50 | 24 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (15.2) | 49.5 (16.5) | 49.2 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 13 | 44
  Male | 19 | 11 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 24 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 50 | 24 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stable Platelet Response of at Least 50,000/µL
Description: Stable platelet response by Week 24 defined as a platelet count of at least 50,000/µL on at least 4 of the 6 visits between Weeks 14-24
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 50 | 24
Participants | 9 | 1
Statistical Analysis 1: Comparison: Fostamatinib Recipient; Test type: Superiority; p = 0.1519, Fisher Exact; Risk Difference (RD) = 13.8, 95% CI 2-sided [0.5 to 27.1] — Confidence interval for treatment difference (risk difference) was based on the normal approximation

2. Secondary Outcome: Number of Participants With Platelet Count ≥ 50,000/µL at Week 12
Description: Platelet Count ≥ 50,000/µL at Week 12
Time Frame: Baseline to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 50 | 24
Participants | 12 | 3

3. Secondary Outcome: Number of Participants With Platelet Count ≥ 50,000/µL at Week 24
Description: Platelet Count ≥ 50,000/µL at Week 24
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 50 | 24
Participants | 8 | 1

4. Secondary Outcome: Number of Participants With Platelet Count ≥ 30,000/μL and at Least 20,000/μL Above Baseline at Week 12
Description: Among subjects with a baseline platelet count < 15,000/μL, achievement of a count ≥ 30,000/μL and at least 20,000/μL above baseline at Week 12.
Time Frame: Baseline to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 22 | 9
Participants | 6 | 1

5. Secondary Outcome: Number of Participants With Platelet Count ≥ 30,000/μL and at Least 20,000/μL Above Baseline at Week 24
Description: Among subjects with a baseline platelet count < 15,000/μL, achievement of a count ≥ 30,000/μL and at least 20,000/μL above baseline at Week 24
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 22 | 9
Participants | 3 | 0

6. Secondary Outcome: Frequency and Severity of Bleeding According to the ITP Bleeding Score (IBLS)
Description: The ITP Bleeding Scale (IBLS) is an immune thrombocytopenic purpura (ITP)-specific bleeding score used to analyze the correlation of clinical and laboratory platelet variables with bleeding. The IBLS comprises of 11 grades from 0 (none) to 2 (marked bleeding) by history over the previous week or by exam; 2 being worse. These 11 grades include: skin by physical exam, oral by physical exam, skin by history, oral by history, epistaxis, gastrointestinal, urinary, gynecological, pulmonary, intracranial hemorrhage, and subconjunctival hemorrhage. After each grade is scored, the mean value for all 11 grades is calculated (lowest score being 0 and highest score being 2) for each subject visit. LOCF method was used to impute any missing data.
  The mean of the IBLS scores across visits during the 24-week treatment period was summarized by treatment group using descriptive statistics. A 2-sided, 2-sample t-test was used to test for a difference in means between treatments for this endpoint.
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 50 | 24
scores on a scale | 0.04 (0.08) | 0.06 (0.07)
Statistical Analysis 1: Comparison: Fostamatinib Recipient vs Placebo Recipient; Test type: Superiority; p = 0.4927, t-test, 2 sided — P-value from a two-sided two-sample t-test, testing for a difference in means between fostamatinib and placebo; Risk Difference (RD) = -0.01, 95% CI 2-sided [-0.05 to 0.02]

7. Secondary Outcome: Frequency and Severity of Bleeding According to the World Health Organization (WHO) Bleeding Scale
Description: The World Health Organization (WHO) bleeding scale is a standardized grading scale created to measure the severity of bleeding. The scale is a clinical investigator-assessed five-point scale with a score range starting at the lowest 0=No bleeding, 1 = Petechiae, 2=Mild blood loss, 3=Gross blood loss, to the worse 4=Debilitating blood loss. The WHO bleeding scale is scored by history over the previous-week or by exam. After each grade is scored, the mean value is calculated (lowest score being 0 [no bleeding] to the highest score being 4 [debilitating blood loss]) for each visit. LOCF method was used to impute any missing data.
  The mean of the WHO bleeding scale across visits during the 24-week treatment period was summarized by treatment group using descriptive statistics. A 2-sided, 2-sample t-test was used to test for a difference in means between treatments for this endpoint.
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 50 | 24
scores on a scale | 0.26 (0.38) | 0.38 (0.47)
Statistical Analysis 1: Comparison: Fostamatinib Recipient vs Placebo Recipient; Test type: Superiority; p = 0.2499, t-test, 2 sided — P-value from a two-sided two-sample t-test, testing for a difference in means between fostamatinib and placebo; Risk Difference (RD) = -0.12, 95% CI 2-sided [-0.32 to 0.09]

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: One patient randomized to the placebo group was given the wrong treatment kit, and was treated with fostamatinib for 2 weeks. This patient's efficacy data were analyzed with the placebo arm, but his safety data were analyzed with the fostamatinib arm.
Arm/Group | Fostamatinib Recipient | Placebo Recipient
All-Cause Mortality (participants affected / at risk) | 1/51 | 0/23
Serious Adverse Events (participants affected / at risk) | 5/51 | 6/23
Other Adverse Events (participants affected / at risk) | 36/51 | 18/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fostamatinib Recipient (N=51) | Placebo Recipient (N=23)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (8)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fostamatinib Recipient (N=51) | Placebo Recipient (N=23)
Diarrhoea (Gastrointestinal disorders) | 9 | 3
Nausea (Gastrointestinal disorders) | 4 | 3
Haematoma (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 7 | 3
Bronchitis (Infections and infestations) | 3 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Headache (Nervous system disorders) | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No